CLINICAL TRIAL: NCT00951769
Title: A Comparison of the Difficult Airway Society (UK) and Australian Patient Safety Foundation Crisis Algorithms for Difficult Intubation in a Simulated Difficult Intubation Scenario
Brief Title: Algorithms in a Simulated Difficult Intubation Scenario
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 09/H1001/3
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2009-08

CONDITIONS: Airway Management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control,: Control
- DAS: Difficult Airway Society, UK: DAS difficult airway algorithm
- Australian: Australian difficult airway algorithm

SUMMARY:
This is a non-human study, conducted in a simulation environment, with simulator manikins, and volunteers from anaesthesia. Trainees in their first 2 years of anaesthetics training will be randomised to a control group, a group following the Difficult Airway Society UK's Guidelines and the Australian Difficult Airway management algorithm. A simulated difficult airway will be created during the induction of anaesthesia. The investigators will examine adherence to guidelines, which would have been provided to participants before the experiment, as well as compare their performance with the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthetists in first 2 years of training

Exclusion Criteria:

* Those who decline invitation to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Trainee anaesthetists in for 2 years of training
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Time to safe oxygenation for manikin | Variable

CONTACTS AND LOCATIONS:
Overall Officials: ARPAN GUHA, MD, FRCA, Principal Investigator — AINTREE HOSPITALS NHS TRUST
Locations (1):
- Cheshire & Merseyside Simulation Centre, Liverpool, Merseyside, United Kingdom